CLINICAL TRIAL: NCT05526716
Title: A Phase 3 Randomized, Double-blind, Placebo-Controlled Clinical Study to Evaluate the Safety, Tolerability, and Immunogenicity of V116 When Administered Concomitantly With Influenza Vaccine in Adults 50 Years of Age or Older
Brief Title: A Study to Evaluate the Safety, Tolerability, and Immunogenicity of V116 When Administered Concomitantly With Influenza Vaccine in Adults 50 Years of Age or Older (V116-005, STRIDE-5)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V116-005
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Pneumonia, Pneumococcal
MeSH Terms: conditions — Pneumonia, Pneumococcal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Concomitant group (V116 + QIV followed by placebo) (Experimental): Participants will receive a single 0.5 mL intramuscular (IM) injection of V116 and a single 0.5 mL IM injection of QIV on Day 1 and a single 0.5 mL injection of placebo on Day 30
  Interventions: Biological: V116; Biological: QIV; Biological: Matching Placebo for V116
- Sequential group (placebo + QIV followed by V116) (Experimental): Participants will receive a single 0.5 mL IM injection of QIV and a single 0.5 mL IM injection of placebo on Day 1 and a single 0.5 mL injection of V116 on Day 30
  Interventions: Biological: V116; Biological: QIV; Biological: Matching Placebo for V116

INTERVENTIONS:
Biological: V116 — Pneumococcal 21-valent conjugate vaccine with 4 μg of each of the pneumococcal polysaccharides (PnPs) antigen: 3, 6A, 7F, 8, 9N, 10A, 11A, 12F, 15A, 15C, 16F, 17F, 19A, 20A, 22F, 23A, 23B, 24F, 31, 33F, and 35B in each 0.5 mL sterile solution
Biological: QIV — Single 0.5 mL IM injection
Biological: Matching Placebo for V116 — Single 0.5 mL of sterile saline IM injection

SUMMARY:
This a study of V116 in adults ≥50 years of age who concomitantly received Influenza vaccine. The primary objectives of this study are to evaluate the safety, tolerability, and immunogenicity of V116 when administered concomitantly with Quadrivalent Influenza Vaccine (QIV) compared with V116 administered sequentially with QIV. The primary hypotheses state that immune responses to V116 and to QIV are non-inferior when administered concomitantly as compared with sequential administration as measured by serotype-specific opsonophagocytic activity (OPA) for V116 and hemagglutination inhibition (HAI) geometric mean titers (GMTs) for QIV, at 30 days postvaccination.

ELIGIBILITY:
Inclusion Criteria:

* Any underlying chronic conditions were assessed to be in stable condition per the investigator's judgment
* Females: Not pregnant or a breast feeding and not a woman of childbearing potential (WOCBP) or a WOCBP agrees to use contraception or remain abstinent

Exclusion Criteria:

* History of IPD or other culture-positive pneumococcal disease
* Known or suspected impairment of immunological function
* Receipt of systemic corticosteroids or immunosuppressive therapy
* Received any pneumococcal vaccine <12 months prior to enrollment
* Prior administration of PCV15 or PCV20
* Received any influenza vaccine <6 months prior to enrollment

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1080 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (56):
- United States (56):
  - Central Phoenix Medical Clinic-Synexus Clinical Research US ( Site 0012), Phoenix, Arizona
  - Hope Clinical Research, Inc. ( Site 0070), Canoga Park, California
  - Paradigm Clinical Research Centers, Inc ( Site 0024), La Mesa, California
  - Catalina Research Institute, LLC ( Site 0067), Montclair, California
  - WR- PRI, LLC ( Site 0044), Newport Beach, California
  - Carbon Health - North Hollywood - NoHo West ( Site 0016), North Hollywood, California
  - Valley Clinical Trials, Inc. ( Site 0002), Northridge, California
  - Artemis Institute for Clinical Research ( Site 0023), San Diego, California
  - WR-MCCR, LLC ( Site 0033), San Diego, California
  - California Research Foundation ( Site 0005), San Diego, California
  - Diablo Clinical Research, Inc. ( Site 0020), Walnut Creek, California
  - Velocity Clinical Research, Hallandale Beach ( Site 0064), Hallandale, Florida
  - Indago Research & Health Center, Inc ( Site 0029), Hialeah, Florida
  - East Coast Institute for Research, LLC ( Site 0013), Jacksonville, Florida
  - Health Awareness ( Site 0034), Jupiter, Florida
  - Optimal Research ( Site 0008), Melbourne, Florida
  - Suncoast Research Group-Clinical Department ( Site 0062), Miami, Florida
  - Suncoast Research Associates ( Site 0041), Miami, Florida
  - Alpha Science Research ( Site 0042), Miami, Florida
  - Lakes Research ( Site 0063), Miami Lakes, Florida
  - Triple O Research Institute, P.A ( Site 0054), West Palm Beach, Florida
  - East Coast Institute for Research - Canton ( Site 0004), Canton, Georgia
  - Clinical Research Atlanta ( Site 0068), Stockbridge, Georgia
  - Synexus Clinical Research US, Inc. ( Site 0072), Chicago, Illinois
  - Healthcare Research Network - Chicago ( Site 0014), Flossmoor, Illinois
  - Centennial Medical Group ( Site 0035), Elkridge, Maryland
  - Healthcare Research Network - St. Louis ( Site 0011), St Louis, Missouri
  - Radiant Research ( Site 0073), St Louis, Missouri
  - Alivation Research-Primary Care ( Site 0066), Lincoln, Nebraska
  - WR-CRCN, LLC ( Site 0018), Las Vegas, Nevada
  - Axces Research ( Site 0037), Santa Fe, New Mexico
  - Smith Allergy and Asthma Specialists-Certified Research Associates ( Site 0019), Cortland, New York
  - Synexus Clinical Research US, Inc - New York ( Site 0053), New York, New York
  - Rochester Clinical Research, Inc. ( Site 0055), Rochester, New York
  - Meridian Clinical Research, LLC ( Site 0032), Vestal, New York
  - Carolina Institute for Clinical Research ( Site 0047), Fayetteville, North Carolina
  - M3 Wake Research Associates ( Site 0040), Raleigh, North Carolina
  - CTI Clinical Research Center ( Site 0071), Cincinnati, Ohio
  - Velocity Clinical Research, Medford ( Site 0060), Medford, Oregon
  - Hatboro Medical Associates / CCT Research ( Site 0065), Hatboro, Pennsylvania
  - Velocity Clinical Research, Providence ( Site 0021), East Greenwich, Rhode Island
  - Velocity Clinical Research, Anderson ( Site 0077), Anderson, South Carolina
  - Velocity Clinical Research, Columbia ( Site 0058), Columbia, South Carolina
  - Holston Medical Group-Clinical Research ( Site 0028), Bristol, Tennessee
  - Holston Medical Group-Clinical Research ( Site 0009), Kingsport, Tennessee
  - Clinical Research Associates Inc ( Site 0026), Nashville, Tennessee
  - Optimal Research ( Site 0015), Austin, Texas
  - Headlands Research - Brownsville ( Site 0069), Brownsville, Texas
  - Benchmark Research ( Site 0025), Fort Worth, Texas
  - New Horizon Medical Group ( Site 0078), Houston, Texas
  - Innovative Medical Research of Texas ( Site 0079), Houston, Texas
  - LinQ Research ( Site 0074), Pearland, Texas
  - Synexus Clinical Research US, Inc. ( Site 0001), Murray, Utah
  - Alliance for Multispecialty Research, LLC ( Site 0051), South Jordan, Utah
  - Arthritis Northwest, PLLC ( Site 0059), Spokane, Washington
  - Velocity Clinical Research, Spokane ( Site 0050), Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Omole T, Weinberg AS, Azizad M, Greenberg D, Grijalva CG, Orenstein WA, Euler D, Fernsler D, Park J, Li J, Platt HL; STRIDE-5 study group. A phase 3 randomized, double-blind clinical study to evaluate the safety and immunogenicity of V116 when administered concomitantly with influenza vaccine in adults 50 years of age or older. Vaccine. 2025 Aug 30;62:127514. doi: 10.1016/j.vaccine.2025.127514. Epub 2025 Jul 25. PMID 40714528
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26087&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 56 centers in the United States.
Groups:
- Concomitant Group (V116 + QIV Followed by Placebo): Participants received a single 0.5 mL intramuscular (IM) injection of V116 and a single 0.5 mL IM injection of quadrivalent influenza vaccine (QIV) on Day 1 and a single 0.5 mL injection of placebo on Day 30.
- Sequential Group (Placebo + QIV Followed by V116): Participants received a single 0.5 mL IM injection of QIV and a single 0.5 mL IM injection of placebo on Day 1 and a single 0.5 mL injection of V116 on Day 30.
Period: Overall Study
Arm/Group | Concomitant Group (V116 + QIV Followed by Placebo) | Sequential Group (Placebo + QIV Followed by V116)
Started | 540 | 540
Vaccinated at Visit 1 (QIV) | 536 | 536
Vaccinated at Visit 1 (V116) | 534 | 0
Vaccinated at Visit 1 (Placebo) | 0 | 535
Vaccinated at Visit 3 (Placebo) | 522 | 0
Vaccinated at Visit 3 (V116) | 0 | 518
Completed | 510 | 507
Not Completed | 30 | 33
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 17 | 15
Not completed — Physician Decision | 0 | 1
Not completed — Randomized by mistake without study treatment | 0 | 1
Not completed — Withdrawal by Subject | 12 | 12
Not completed — Not reported | 0 | 2

BASELINE CHARACTERISTICS:
Population: All vaccinated participants are included.
Groups:
- Concomitant Group (V116 + QIV Followed by Placebo): Participants received a single 0.5 mL IM injection of V116 and a single 0.5 mL IM injection of QIV on Day 1 and a single 0.5 mL injection of placebo on Day 30.
- Total: Total of all reporting groups
Arm/Group | Concomitant Group (V116 + QIV Followed by Placebo) | Sequential Group (Placebo + QIV Followed by V116) | Total
Number analyzed (Participants) | 536 | 536 | 1072
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (8.4) | 64.2 (8.4) | 64.2 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 297 | 287 | 584
  Male | 239 | 249 | 488
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 127 | 125 | 252
  Not Hispanic or Latino | 403 | 409 | 812
  Unknown or Not Reported | 6 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 4 | 5
  Asian | 3 | 10 | 13
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 107 | 101 | 208
  White | 410 | 412 | 822
  More than one race | 13 | 8 | 21
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Injection-site Adverse Events (AEs)
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited injection-site AEs included erythema, pain, and swelling.
Time Frame: Up to 5 days post-vaccination
Population: All randomized participants who received at least 1 dose of study vaccination and received QIV are included, according to actual vaccination received.
Measure: Count of Participants; unit: Participants
Arm/Group | Concomitant Group (V116 + QIV Followed by Placebo) | Sequential Group (Placebo + QIV Followed by V116)
Number analyzed (Participants) | 534 | 535
Participants | 317 | 314

2. Primary Outcome: Number of Participants With Solicited Systemic AEs
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Solicited systemic AEs include fatigue, headache, myalgia, and pyrexia.
Time Frame: Up to 5 days post-vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Concomitant Group (V116 + QIV Followed by Placebo) | Sequential Group (Placebo + QIV Followed by V116)
Number analyzed (Participants) | 534 | 535
Participants | 219 | 224

3. Primary Outcome: Percentage of Participants With Vaccine-related Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires inpatient hospitalization or prolongs existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is another important medical event. SAEs that were reported to be at least possibly related by the investigator to study vaccination are summarized.
Time Frame: Up to ~6 months postvaccination with V116
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Concomitant Group (V116 + QIV Followed by Placebo) | Sequential Group (Placebo + QIV Followed by V116)
Number analyzed (Participants) | 534 | 535
Participants | 0 | 1

4. Primary Outcome: Geometric Mean Titer (GMT) of Serotype-specific Opsonophagocytic Activity (OPA) Responses
Description: OPA for the serotypes in V116 were determined using a multiplexed opsonophagocytic assay (MOPA). Serotype-specific OPA GMTs (GMTs) (estimated) and GMT ratios with 95% CIs were calculated using a constrained longitudinal data analysis (cLDA) model utilizing data from both vaccination groups. Per the statistical analysis plan, the only CIs calculated were the between-group CIs (for the GMT ratios); within-group CIs were not calculated.
Time Frame: 30 days after V116 vaccination (Day 30 for concomitant group and Day 59 for sequential group)
Population: All randomized participants without deviations from the protocol that may substantially affect immunogenicity. Overall participants analyzed were the number of participants randomized and vaccinated with available serotype data; number analyzed for each serotype is the subset of those overall participants analyzed without protocol deviation and with data available for the respective serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Concomitant Group (V116 + QIV Followed by Placebo) | Sequential Group (Placebo + QIV Followed by V116)
Number analyzed (Participants) | 536 | 536
Titers
  3: number analyzed (Participants) | 519 | 497
  3 | 209.2 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 250.1 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  6A: number analyzed (Participants) | 521 | 496
  6A | 2056.4 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 2608.2 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  7F: number analyzed (Participants) | 521 | 496
  7F | 2399.2 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 3275.4 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  8: number analyzed (Participants) | 519 | 497
  8 | 1508.9 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 2135.7 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  9N: number analyzed (Participants) | 522 | 499
  9N | 5075.6 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 7566.6 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  10A: number analyzed (Participants) | 524 | 499
  10A | 3033.6 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 3966.2 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  11A: number analyzed (Participants) | 519 | 499
  11A | 2576.3 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 4051.1 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  12F: number analyzed (Participants) | 525 | 499
  12F | 1869.9 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 2449.5 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  15A: number analyzed (Participants) | 511 | 458
  15A | 4670.6 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 6559.7 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  15C: number analyzed (Participants) | 522 | 493
  15C | 3426.0 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 4832.6 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  16F: number analyzed (Participants) | 522 | 498
  16F | 5371.5 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 7757.2 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  17F: number analyzed (Participants) | 520 | 497
  17F | 5783.8 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 7924.3 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  19A: number analyzed (Participants) | 524 | 498
  19A | 1830.1 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 2453.3 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  20A: number analyzed (Participants) | 522 | 498
  20A | 5172.8 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 6986.9 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  22F: number analyzed (Participants) | 517 | 490
  22F | 3194.9 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 4158.2 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  23A: number analyzed (Participants) | 511 | 486
  23A | 3358.2 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 4319.9 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  23B: number analyzed (Participants) | 522 | 498
  23B | 934.3 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 1664.5 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  24F: number analyzed (Participants) | 517 | 494
  24F | 2996.5 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 4143.1 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  31: number analyzed (Participants) | 522 | 499
  31 | 2997.4 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 4390.6 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  33F: number analyzed (Participants) | 520 | 492
  33F | 9032.5 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 10765.1 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  35B: number analyzed (Participants) | 522 | 495
  35B | 7701.4 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 9940.2 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
Statistical Analysis 1: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); The concomitant group will be considered noninferior to the sequential group if the lower bound of the 2-sided 95% CI of the OPA GMT ratio (GMTcon/GMTseq) for each of the serotypes is >0.50; Test type: Non-Inferiority — Serotype 3; Geometric Mean Titers Ratio (GMT Ratio) = 0.84, 95% CI 2-sided [0.72 to 0.97]
Statistical Analysis 2: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority — Serotype 6A; GMT Ratio = 0.79, 95% CI 2-sided [0.66 to 0.94]
Statistical Analysis 3: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority — Serotype 7F; GMT Ratio = 0.73, 95% CI 2-sided [0.63 to 0.85]
Statistical Analysis 4: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority — Serotype 8; GMT Ratio = 0.71, 95% CI 2-sided [0.61 to 0.82]
Statistical Analysis 5: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority — Serotype 9N; GMT Ratio = 0.67, 95% CI 2-sided [0.57 to 0.79]
Statistical Analysis 6: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority — Serotype 10A; GMT Ratio = 0.76, 95% CI 2-sided [0.65 to 0.91]
Statistical Analysis 7: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority — Serotype 11A; GMT Ratio = 0.64, 95% CI 2-sided [0.54 to 0.75]
Statistical Analysis 8: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority — Serotype 12F; GMT Ratio = 0.76, 95% CI 2-sided [0.62 to 0.94]
Statistical Analysis 9: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority — Serotype 15A; GMT Ratio = 0.71, 95% CI 2-sided [0.60 to 0.85]
Statistical Analysis 10: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority — Serotype 15C; GMT Ratio = 0.71, 95% CI 2-sided [0.58 to 0.87]
Statistical Analysis 11: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority — Serotype 16F; GMT Ratio = 0.69, 95% CI 2-sided [0.59 to 0.81]
Statistical Analysis 12: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority — Serotype 17F; GMT Ratio = 0.73, 95% CI 2-sided [0.62 to 0.86]
Statistical Analysis 13: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority — Serotype 19A; GMT Ratio = 0.75, 95% CI 2-sided [0.65 to 0.85]
Statistical Analysis 14: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority — Serotype 20A; GMT Ratio = 0.74, 95% CI 2-sided [0.63 to 0.87]
Statistical Analysis 15: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority — Serotype 22F; GMT Ratio = 0.77, 95% CI 2-sided [0.65 to 0.91]
Statistical Analysis 16: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority — Serotype 23A; GMT Ratio = 0.78, 95% CI 2-sided [0.63 to 0.96]
Statistical Analysis 17: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority — Serotype 23B; GMT Ratio = 0.56, 95% CI 2-sided [0.44 to 0.72]
Statistical Analysis 18: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority — Serotype 24F; GMT Ratio = 0.72, 95% CI 2-sided [0.61 to 0.86]
Statistical Analysis 19: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority — Serotype 31; GMT Ratio = 0.68, 95% CI 2-sided [0.56 to 0.83]
Statistical Analysis 20: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); [analysis description as in outcome 4, analysis 1]; Test type: Non-Inferiority — Serotype 33F; GMT Ratio = 0.84, 95% CI 2-sided [0.70 to 1.01]
Statistical Analysis 21: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); The concomitant group will be considered noninferior to the sequential group if the lower bound of the 2-sided 95% CI of the OPA GMT ratio (GMTcon/GMTseq) for each of serotypes is >0.50; Test type: Non-Inferiority — Serotype 35B; GMT Ratio = 0.77, 95% CI 2-sided [0.67 to 0.89]

5. Primary Outcome: GMT of Influenza Strain-specific Hemagglutination Inhibition (HAI)
Description: GMTs for the 4 strains contained in QIV vaccine were determined using an HAI assay.
Time Frame: Day 30
Population: All randomized participants without deviations from the protocol that may substantially affect immunogenicity. Deviations include, but are not limited to the following: missing serology results; and blood draw out of window.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Concomitant Group (V116 + QIV Followed by Placebo) | Sequential Group (Placebo + QIV Followed by V116)
Number analyzed (Participants) | 536 | 536
Titers
  A/H1N1 | 268.23 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 325.06 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  A/H3N2 | 128.07 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 163.06 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  B/Victoria | 70.02 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 85.66 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  B/Yamagata | 31.80 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 35.86 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
Statistical Analysis 1: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); The concomitant group will be considered noninferior to the sequential group if the lower bound of the 2-sided 95% CI of the HAI GMT ratio (GMTcon/GMTseq) for each of the strains is >0.67; Test type: Non-Inferiority — A/H1N1; GMT Ratio = 0.83, 95% CI 2-sided [0.70 to 0.97]
Statistical Analysis 2: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); [analysis description as in outcome 5, analysis 1]; Test type: Non-Inferiority — A/H3N2; GMT Ratio = 0.79, 95% CI 2-sided [0.67 to 0.93]
Statistical Analysis 3: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); [analysis description as in outcome 5, analysis 1]; Test type: Non-Inferiority — B/Victoria; GMT Ratio = 0.82, 95% CI 2-sided [0.70 to 0.95]
Statistical Analysis 4: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); [analysis description as in outcome 5, analysis 1]; Test type: Non-Inferiority — B/Yamagata; GMT Ratio = 0.89, 95% CI 2-sided [0.78 to 1.00]

6. Secondary Outcome: Geometric Mean Concentration (GMC) of Serotype-specific Immunoglobulin G (IgG)
Description: The GMCs of serotype-specific IgG for the serotypes contained in V116 were determined using a pneumococcal electrochemiluminescence (Pn ECL) assay.
Time Frame: 30 days after V116 vaccination (Day 30 for concomitant group and Day 59 for sequential group)
Population: All randomized participants without protocol deviations that may substantially affect the results of theimmunogenicity endpoint are included. Overall participants analyzed were the number of participantsrandomized and vaccinated with available serotype data; number analyzed for each serotype is the subset of those overall participants analyzed without protocol deviation and with data available forthe respective serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Concomitant Group (V116 + QIV Followed by Placebo) | Sequential Group (Placebo + QIV Followed by V116)
Number analyzed (Participants) | 536 | 536
µg/mL
  3: number analyzed (Participants) | 528 | 505
  3 | 0.60 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 0.66 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  6A: number analyzed (Participants) | 528 | 505
  6A | 3.34 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 3.58 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  7F: number analyzed (Participants) | 528 | 505
  7F | 3.91 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 5.01 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  8: number analyzed (Participants) | 528 | 505
  8 | 6.84 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 8.38 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  9N: number analyzed (Participants) | 528 | 505
  9N | 4.99 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 5.64 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  10A: number analyzed (Participants) | 528 | 505
  10A | 8.45 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 10.70 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  11A: number analyzed (Participants) | 528 | 505
  11A | 4.83 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 5.84 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  12F: number analyzed (Participants) | 528 | 505
  12F | 1.10 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 1.31 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  15A: number analyzed (Participants) | 528 | 505
  15A | 8.83 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 11.77 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  15C: number analyzed (Participants) | 528 | 505
  15C | 7.13 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 8.39 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  16F: number analyzed (Participants) | 528 | 505
  16F | 1.93 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 2.32 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  17F: number analyzed (Participants) | 528 | 505
  17F | 9.69 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 11.44 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  19A: number analyzed (Participants) | 528 | 504
  19A | 6.41 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 7.91 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  20A: number analyzed (Participants) | 528 | 505
  20A | 13.57 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 16.52 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  22F: number analyzed (Participants) | 528 | 505
  22F | 3.13 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 3.34 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  23A: number analyzed (Participants) | 528 | 505
  23A | 3.30 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 3.87 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  23B: number analyzed (Participants) | 528 | 505
  23B | 4.24 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 4.94 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  24F: number analyzed (Participants) | 528 | 505
  24F | 5.72 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 6.71 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  31: number analyzed (Participants) | 528 | 505
  31 | 2.50 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 2.96 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  33F: number analyzed (Participants) | 528 | 505
  33F | 9.09 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 11.26 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
  35B: number analyzed (Participants) | 528 | 505
  35B | 15.73 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined. | 18.57 [NA to NA] — Per protocol, within group CIs, or any other measures of dispersion, were not determined.
Statistical Analysis 1: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); Test type: Other — Serotype 3; GMC Ratio = 0.90, 95% CI 2-sided [0.80 to 1.02]
Statistical Analysis 2: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); Test type: Other — Serotype 6A; GMC Ratio = 0.93, 95% CI 2-sided [0.79 to 1.11]
Statistical Analysis 3: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); Test type: Other — Serotype 7F; GMC Ratio = 0.78, 95% CI 2-sided [0.67 to 0.90]
Statistical Analysis 4: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); Test type: Other — Serotype 8; GMC Ratio = 0.82, 95% CI 2-sided [0.70 to 0.95]
Statistical Analysis 5: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); Test type: Other — Serotype 9N; GMC Ratio = 0.88, 95% CI 2-sided [0.75 to 1.05]
Statistical Analysis 6: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); Test type: Other — Serotype 10A; GMC Ratio = 0.79, 95% CI 2-sided [0.67 to 0.94]
Statistical Analysis 7: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); Test type: Other — Serotype 11A; GMC Ratio = 0.83, 95% CI 2-sided [0.72 to 0.96]
Statistical Analysis 8: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); Test type: Other — Serotype 12F; GMC Ratio = 0.83, 95% CI 2-sided [0.69 to 1.01]
Statistical Analysis 9: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); Test type: Other — Serotype 15A; GMC Ratio = 0.75, 95% CI 2-sided [0.63 to 0.90]
Statistical Analysis 10: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); Test type: Other — Serotype 15C; GMC Ratio = 0.85, 95% CI 2-sided [0.71 to 1.02]
Statistical Analysis 11: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); Test type: Other — Serotype 16F; GMC Ratio = 0.83, 95% CI 2-sided [0.70 to 0.99]
Statistical Analysis 12: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); Test type: Other — Serotype 17F; GMC Ratio = 0.85, 95% CI 2-sided [0.72 to 0.99]
Statistical Analysis 13: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); Test type: Other — Serotype 19A; GMC Ratio = 0.81, 95% CI 2-sided [0.71 to 0.93]
Statistical Analysis 14: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); Test type: Other — Serotype 20A; GMC Ratio = 0.82, 95% CI 2-sided [0.70 to 0.97]
Statistical Analysis 15: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); Test type: Other — Serotype 22F; GMC Ratio = 0.94, 95% CI 2-sided [0.80 to 1.10]
Statistical Analysis 16: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); Test type: Other — Serotype 23A; GMC Ratio = 0.85, 95% CI 2-sided [0.70 to 1.03]
Statistical Analysis 17: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); Test type: Other — Serotype 23B; GMC Ratio = 0.86, 95% CI 2-sided [0.72 to 1.02]
Statistical Analysis 18: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); Test type: Other — Serotype 24F; GMC Ratio = 0.85, 95% CI 2-sided [0.69 to 1.05]
Statistical Analysis 19: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); Test type: Other — Serotype 31; GMC Ratio = 0.84, 95% CI 2-sided [0.72 to 0.99]
Statistical Analysis 20: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); Test type: Other — Serotype 33F; GMC Ratio = 0.81, 95% CI 2-sided [0.69 to 0.94]
Statistical Analysis 21: Comparison: Concomitant Group (V116 + QIV Followed by Placebo) vs Sequential Group (Placebo + QIV Followed by V116); Test type: Other — Serotype 35B; GMC Ratio = 0.85, 95% CI 2-sided [0.72 to 0.99]

7. Secondary Outcome: Geometric Mean Fold Rise (GMFR) Ratio of Serotype-specific OPA
Description: OPA for the serotypes in V116 were determined using a MOPA. GMFR ratio is defined as the geometric mean of the ratio of concentration at Day 30 after vaccination divided by concentration at baseline.
Time Frame: Baseline (Day 1 for the concomitant group and Day 30 for the sequential group) and Postvaccination (Day 30 for the concomitant group and Day 59 for the sequential group)
Population: All randomized participants without protocol deviations that may substantially affect the results of the immunogenicity endpoint and have all data available are included. Overall participants analyzed were the number of participants randomized and vaccinated with available serotype data; number analyzed for each serotype is the subset of those overall participants analyzed without protocol deviation and with data available for the respective serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Concomitant Group (V116 + QIV Followed by Placebo) | Sequential Group (Placebo + QIV Followed by V116)
Number analyzed (Participants) | 536 | 536
Ratio
  3: number analyzed (Participants) | 427 | 403
  3 | 5.2 [4.6 to 5.9] | 6.7 [5.9 to 7.6]
  6A: number analyzed (Participants) | 430 | 400
  6A | 9.4 [8.0 to 11.1] | 13.2 [11.0 to 15.8]
  7F: number analyzed (Participants) | 451 | 395
  7F | 8.1 [6.8 to 9.6] | 9.8 [8.1 to 11.9]
  8: number analyzed (Participants) | 457 | 420
  8 | 9.6 [8.0 to 11.6] | 10.9 [9.0 to 13.3]
  9N: number analyzed (Participants) | 452 | 408
  9N | 6.2 [5.3 to 7.4] | 8.2 [6.9 to 9.6]
  10A: number analyzed (Participants) | 459 | 429
  10A | 10.4 [8.7 to 12.6] | 11.1 [9.2 to 13.4]
  11A: number analyzed (Participants) | 435 | 395
  11A | 13.0 [10.7 to 15.9] | 15.2 [12.4 to 18.7]
  12F: number analyzed (Participants) | 463 | 429
  12F | 37.4 [30.8 to 45.5] | 46.8 [37.7 to 58.0]
  15A: number analyzed (Participants) | 344 | 269
  15A | 7.6 [6.4 to 9.1] | 8.9 [7.3 to 11.0]
  15C: number analyzed (Participants) | 447 | 411
  15C | 25.0 [20.5 to 30.4] | 30.2 [24.5 to 37.3]
  16F: number analyzed (Participants) | 436 | 397
  16F | 9.9 [8.6 to 11.4] | 11.9 [10.3 to 13.7]
  17F: number analyzed (Participants) | 455 | 405
  17F | 10.4 [8.8 to 12.4] | 15.1 [12.8 to 18.0]
  19A: number analyzed (Participants) | 463 | 422
  19A | 3.6 [3.2 to 4.2] | 5.2 [4.5 to 6.1]
  20A: number analyzed (Participants) | 444 | 397
  20A | 6.7 [5.7 to 7.7] | 8.5 [7.3 to 9.9]
  22F: number analyzed (Participants) | 443 | 390
  22F | 13.7 [11.2 to 16.8] | 16.9 [13.6 to 20.9]
  23A: number analyzed (Participants) | 367 | 339
  23A | 17.0 [14.0 to 20.8] | 25.5 [20.4 to 31.8]
  23B: number analyzed (Participants) | 460 | 417
  23B | 42.9 [35.4 to 52.0] | 60.9 [48.9 to 75.9]
  24F: number analyzed (Participants) | 403 | 376
  24F | 31.6 [26.1 to 38.3] | 33.2 [27.3 to 40.5]
  31: number analyzed (Participants) | 432 | 392
  31 | 29.8 [24.5 to 36.2] | 40.3 [32.5 to 49.9]
  33F: number analyzed (Participants) | 409 | 377
  33F | 5.5 [4.7 to 6.4] | 6.3 [5.3 to 7.4]
  35B: number analyzed (Participants) | 409 | 377
  35B | 5.5 [4.7 to 6.4] | 6.3 [5.3 to 7.4]

8. Secondary Outcome: GMFR Ratio of Serotype-specific IgG
Description: GMFR ratios for the serotype-specific IgG in V116 were determined using a Pn ECL.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Concomitant Group (V116 + QIV Followed by Placebo) | Sequential Group (Placebo + QIV Followed by V116)
Number analyzed (Participants) | 536 | 536
Ratio
  3: number analyzed (Participants) | 493 | 457
  3 | 3.6 [3.3 to 4.0] | 4.1 [3.7 to 4.6]
  6A: number analyzed (Participants) | 493 | 457
  6A | 7.8 [6.9 to 8.9] | 8.4 [7.3 to 9.7]
  7F: number analyzed (Participants) | 493 | 459
  7F | 5.6 [5.0 to 6.4] | 7.2 [6.3 to 8.2]
  8: number analyzed (Participants) | 493 | 459
  8 | 7.1 [6.2 to 8.1] | 8.7 [7.5 to 10.1]
  9N: number analyzed (Participants) | 493 | 458
  9N | 8.0 [6.9 to 9.2] | 9.0 [7.8 to 10.5]
  10A: number analyzed (Participants) | 493 | 457
  10A | 9.3 [8.1 to 10.6] | 11.4 [9.9 to 13.1]
  11A: number analyzed (Participants) | 493 | 459
  11A | 5.7 [5.1 to 6.4] | 7.2 [6.3 to 8.1]
  12F: number analyzed (Participants) | 493 | 459
  12F | 6.9 [6.0 to 8.0] | 7.9 [6.8 to 9.1]
  15A: number analyzed (Participants) | 493 | 458
  15A | 14.2 [12.3 to 16.4] | 19.5 [16.8 to 22.5]
  15C: number analyzed (Participants) | 493 | 458
  15C | 11.0 [9.6 to 12.6] | 12.3 [10.6 to 14.2]
  16F: number analyzed (Participants) | 493 | 458
  16F | 11.1 [9.8 to 12.6] | 13.4 [11.8 to 15.2]
  17F: number analyzed (Participants) | 493 | 459
  17F | 10.9 [9.5 to 12.5] | 13.2 [11.5 to 15.3]
  19A: number analyzed (Participants) | 493 | 458
  19A | 3.0 [2.7 to 3.4] | 3.9 [3.5 to 4.5]
  20A: number analyzed (Participants) | 493 | 459
  20A | 7.4 [6.5 to 8.4] | 8.9 [7.7 to 10.2]
  22F: number analyzed (Participants) | 493 | 459
  22F | 8.2 [7.1 to 9.4] | 9.0 [7.8 to 10.3]
  23A: number analyzed (Participants) | 493 | 459
  23A | 15.5 [13.6 to 17.6] | 17.3 [15.0 to 20.0]
  23B: number analyzed (Participants) | 493 | 459
  23B | 10.2 [8.9 to 11.6] | 10.9 [9.4 to 12.6]
  24F: number analyzed (Participants) | 493 | 459
  24F | 20.2 [17.4 to 23.4] | 23.5 [20.3 to 27.3]
  31: number analyzed (Participants) | 493 | 459
  31 | 12.6 [11.2 to 14.2] | 15.3 [13.5 to 17.3]
  33F: number analyzed (Participants) | 493 | 459
  33F | 5.1 [4.5 to 5.7] | 6.2 [5.4 to 7.1]
  35B: number analyzed (Participants) | 493 | 458
  35B | 12.3 [10.9 to 13.9] | 14.9 [13.0 to 17.1]

9. Secondary Outcome: GMFR in Influenza Strain-specific HAI
Description: Activity for the 4 strains contained in QIV vaccine was determined using an HAI assay. GMFR is GMT 30 days after vaccination / GMT at Baseline.
Time Frame: Day 1 (Baseline) and Day 30 (Postvaccination)
Population: All randomized participants without deviations from the protocol that may substantially affect immunogenicity, and who have both baseline and Day 30 data, are included. Deviations include, but are not limited to the following: missing serology results; and blood draw out of window.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Concomitant Group (V116 + QIV Followed by Placebo) | Sequential Group (Placebo + QIV Followed by V116)
Number analyzed (Participants) | 484 | 482
Ratio
  A/H1N1 | 4.5 [3.9 to 5.2] | 5.7 [4.9 to 6.7]
  A/H3N2 | 5.6 [5.0 to 6.3] | 7.1 [6.3 to 8.1]
  B/Victoria | 3.6 [3.3 to 4.0] | 4.5 [4.0 to 5.1]
  B/Yamagata | 1.9 [1.8 to 2.1] | 2.2 [2.1 to 2.4]

10. Secondary Outcome: Percentage of Participants Who Seroconvert for Influenza Strain-specific HAI Titer ≥1:40
Description: The percentage of participants with seroconversion is presented. Activity for the 4 strains contained in QIV vaccine was determined using an HAI assay.
Time Frame: Day 30
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Concomitant Group (V116 + QIV Followed by Placebo) | Sequential Group (Placebo + QIV Followed by V116)
Number analyzed (Participants) | 484 | 482
Percentage of Participants
  A/H1N1 | 47.1 [42.6 to 51.7] | 55.6 [51.0 to 60.1]
  A/H3N2 | 63.8 [59.4 to 68.1] | 68.3 [63.9 to 72.4]
  B/Victoria | 52.3 [47.7 to 56.8] | 54.1 [49.6 to 58.7]
  B/Yamagata | 23.3 [19.6 to 27.4] | 29.9 [25.8 to 34.2]

ADVERSE EVENTS:
Time Frame: Up to ~6 months postvaccination with V116
Description: All-cause mortality is assessed in all randomized participants. Adverse events (AEs) and serious adverse events (SAEs) are reported for all participants as treated.
Arm/Group | Concomitant Group (V116 + QIV Followed by Placebo) | Sequential Group (Placebo + QIV Followed by V116)
All-Cause Mortality (participants affected / at risk) | 1/540 | 2/540
Serious Adverse Events (participants affected / at risk) | 10/534 | 17/535
Other Adverse Events (participants affected / at risk) | 362/534 | 348/535
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concomitant Group (V116 + QIV Followed by Placebo) (N=534) | Sequential Group (Placebo + QIV Followed by V116) (N=535)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Complicated appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Douglas' abscess (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Scrotal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Benign fallopian tube neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Victim of homicide (Social circumstances) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concomitant Group (V116 + QIV Followed by Placebo) (N=534) | Sequential Group (Placebo + QIV Followed by V116) (N=535)
Fatigue (General disorders) | 162 (191) | 175 (218)
Injection site erythema (General disorders) | 63 (75) | 60 (68)
Injection site pain (General disorders) | 310 (481) | 303 (465)
Injection site swelling (General disorders) | 68 (83) | 66 (74)
Myalgia (Musculoskeletal and connective tissue disorders) | 74 (79) | 80 (86)
Headache (Nervous system disorders) | 109 (128) | 120 (142)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/16/NCT05526716/Prot_SAP_000.pdf